CLINICAL TRIAL: NCT01815437
Title: Evaluation of Vitamin D in a Mushroom Supplement
Brief Title: Evaluating Vitamin D Content in Mushrooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MU100
Record Dates: First submitted 2012-02-02; First posted 2013-03-21 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2000 IU Vitamin D3- Cholecalciferol (Active Comparator): Take 2000 IU crystalline vitamin D3 once/day for 12 weeks.
  Interventions: Dietary Supplement: Cholecalciferol
- 2000 IU Vitamin D2- Ergocalciferol (Active Comparator): Take 2000 IU crystalline vitamin D2 supplement once/day for 12 weeks.
  Interventions: Dietary Supplement: Vitamin D2 - Ergocalciferol
- 2000 IU Mushroom Vitamin D2 (Experimental): Take 2000 IU vitamin D2 in a mushroom supplement once/day for 12 weeks
  Interventions: Dietary Supplement: Mushroom Vitamin D2
- Mushroom Extract (Placebo Comparator): Capsules with mushroom extract and no vitamin D. The intervention is mushroom extract.
  Interventions: Dietary Supplement: Mushroom Extract

INTERVENTIONS:
Dietary Supplement: Mushroom Vitamin D2 — 2000 IU vitamin D2 in a mushroom extract, once/day for 12 weeks
  Other Names: Ergocalciferol
  Arms: 2000 IU Mushroom Vitamin D2
Dietary Supplement: Cholecalciferol — 2000 IU crystalline cholecalciferol once/day for 12 weeks
  Arms: 2000 IU Vitamin D3- Cholecalciferol
Dietary Supplement: Vitamin D2 - Ergocalciferol — 2000 IU vitamin D2, ergocalciferol once/day for 12 weeks
  Other Names: Ercocalciferol
  Arms: 2000 IU Vitamin D2- Ergocalciferol
Dietary Supplement: Mushroom Extract — Same quantity of mushroom extract in a capsule
  Arms: Mushroom Extract

SUMMARY:
This study will evaluate how much vitamin D is present in a mushroom supplement. This supplement contains an extract from mushrooms that have been exposed to sunlight. The mushroom supplement will be compared to non-commercially available vitamin D supplements produced in a Goo Manufacturing Practices (GMP)-licensed facility.

DETAILED DESCRIPTION:
Mushrooms have the capability to produce vitamin D in a similar way to human skin. When exposed to ultraviolet light, mushrooms will convert a precursor to vitamin D. This reaction produces large amounts of vitamin D. This study is comparing a natural source of vitamin D to a synthetic source of vitamin D and will help determine if mushrooms are a novel source for this essential nutrient.

ELIGIBILITY:
Inclusion Criteria:

* All healthy adults, male and female, age 18-64 years

Exclusion Criteria:

* Currently taking, or having taken less than one month prior to start of study, a prescription of 50,000 IU of vitamin D2 or 2000 IU vitamin D2 or vitamin D3
* Allergy to mushrooms
* History of elevated calcium (>10.4 mg%)
* Patients with a current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
* Supplementation with over the counter formulations of vitamin D2 or vitamin D3
* Subjects with a history of an adverse reaction to orally administered vitamin D.
* Subjects who are taking oral Dilantin or glucocorticoids.
* Exposure to a tanning bed or tanning on a beach for more than eight hours with no sunscreen within 2 weeks prior to start of study.
* History of intestinal malabsorption (i.e. cystic fibrosis, fat malabsorption syndrome, Crohn's Disease, gastric bypass surgery).
* Subjects with any other condition which in the Investigator's judgment would make the patient unsuitable for inclusion in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in total 25(OH)D in mushroom supplement or crystalline supplement | 12 weeks
  The primary outcome of this study is to examine changes in total 25(OH)D levels after ingestion of a vitamin D2 mushroom supplement manufactured by Monterey Mushrooms, Inc. compared to crystalline vitamin D2 from Nature's Life or vitamin D3 manufactured by Whole Health, Inc.

SECONDARY OUTCOMES:
Changes in gene expression due to mushroom supplement or crystalline supplement | 12 weeks
  The secondary outcome is to look at changes in gene expression, specifically if ingestion of 2000 IU vitamin D2 in a dried mushroom extract and the same quantity of mushroom extract once/day for three months has any added benefits or differences compared to taking crystalline vitamin D2 or vitamin D3.

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, PhD, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Rovner AJ, O'Brien KO. Hypovitaminosis D among healthy children in the United States: a review of the current evidence. Arch Pediatr Adolesc Med. 2008 Jun;162(6):513-9. doi: 10.1001/archpedi.162.6.513. PMID 18524740
- [Background] Kumar J, Muntner P, Kaskel FJ, Hailpern SM, Melamed ML. Prevalence and associations of 25-hydroxyvitamin D deficiency in US children: NHANES 2001-2004. Pediatrics. 2009 Sep;124(3):e362-70. doi: 10.1542/peds.2009-0051. Epub 2009 Aug 3. PMID 19661054
- [Background] Looker AC, Pfeiffer CM, Lacher DA, Schleicher RL, Picciano MF, Yetley EA. Serum 25-hydroxyvitamin D status of the US population: 1988-1994 compared with 2000-2004. Am J Clin Nutr. 2008 Dec;88(6):1519-27. doi: 10.3945/ajcn.2008.26182. PMID 19064511
- [Background] Liu PT, Stenger S, Li H, Wenzel L, Tan BH, Krutzik SR, Ochoa MT, Schauber J, Wu K, Meinken C, Kamen DL, Wagner M, Bals R, Steinmeyer A, Zugel U, Gallo RL, Eisenberg D, Hewison M, Hollis BW, Adams JS, Bloom BR, Modlin RL. Toll-like receptor triggering of a vitamin D-mediated human antimicrobial response. Science. 2006 Mar 24;311(5768):1770-3. doi: 10.1126/science.1123933. Epub 2006 Feb 23. PMID 16497887
- [Background] Ginde AA, Mansbach JM, Camargo CA Jr. Association between serum 25-hydroxyvitamin D level and upper respiratory tract infection in the Third National Health and Nutrition Examination Survey. Arch Intern Med. 2009 Feb 23;169(4):384-90. doi: 10.1001/archinternmed.2008.560. PMID 19237723
- [Background] Holick MF, Biancuzzo RM, Chen TC, Klein EK, Young A, Bibuld D, Reitz R, Salameh W, Ameri A, Tannenbaum AD. Vitamin D2 is as effective as vitamin D3 in maintaining circulating concentrations of 25-hydroxyvitamin D. J Clin Endocrinol Metab. 2008 Mar;93(3):677-81. doi: 10.1210/jc.2007-2308. Epub 2007 Dec 18. PMID 18089691
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] Pietras SM, Obayan BK, Cai MH, Holick MF. Vitamin D2 treatment for vitamin D deficiency and insufficiency for up to 6 years. Arch Intern Med. 2009 Oct 26;169(19):1806-8. doi: 10.1001/archinternmed.2009.361. No abstract available. PMID 19858440